CLINICAL TRIAL: NCT02247869
Title: Dose-dense ABVD as First Line Therapy in Early Stage Unfavorable Hodgkin's Lymphoma: a Phase II, Prospective, Multi-center Study
Brief Title: Dose-dense ABVD First Line Therapy in Early Stage Unfavorable Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL - DDABVD
Record Dates: First submitted 2014-03-07; First posted 2014-09-25 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Hodgkin Lymphoma
Keywords: HL; Hodgkin Lymphoma; First line therapy
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dose dense ABVD (Experimental): 1 arm for all patients (dose dense ABVD on day 1 and 8 every 21 days)
  Interventions: Drug: dose dense ABVD

INTERVENTIONS:
Drug: dose dense ABVD — dose dense ABVD will be administered intravenously on day 1 and 8 every 21 days Chemotherapy regimen
  * Doxorubicin 25 mg/m2 i.v. day 1 and 8
  * Bleomycin 10 mg/m2 i.v. day 1 and 8
  * Vinblastine 6 mg/m2 i.v. day 1 and 8
  * Dacarbazine 375 mg/m2 i.v. day 1 and 8
  Granulocyte colony-stimulating factor (G-CSF): days 9 to 14

SUMMARY:
Prospective, multicenter, Phase II trial designed to assess whether intensification of ABVD (dd-ABVD) is feasible and can improve the outcome of patients with early stage Hodgkin Lymphoma.

DETAILED DESCRIPTION:
Dose-density has been shown to be an important factor for complete remission rate and longterm survival in lymphomas.

The aims of this study were to find out whether intensification of ABVD (dd-ABVD) is feasible and can improve the outcome of patients with early stage Hodgkin Lymphoma. In view of emerging data on the role of early PET in defining prognosis in Hodgkin Lymphoma patients, the percentage of FDG-PET (fluorodeoxyglucose positron emission tomography) negativity after two cycle was chosen as the parameter to evaluate dd-ABVD activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Histologically confirmed Hodgkin Lymphoma stage I, II unfavorable according to EORTC (European Organisation for Research and Treatment of Cancer) criteria, with exclusion of stage II B bulky.
* Previously untreated
* ECOG (Eastern Cooperative Oncology Group) performance status 0 - 2
* Staging with FDG-PET (fluorodeoxyglucose positron emission tomography)
* Written informed consent
* Adequate liver and renal function (total serum bilirubin < 2.5 x ULN, AST/SGOT and/or ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement, serum creatinine < 2.5 x ULN)

Exclusion Criteria:

* Concomitant cardiac, pulmonary, neurologic, psychiatric or metabolic severe disease.
* Uncontrolled diabetes mellitus (with fasting glucose levels above 200mg/dl)
* Other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast or other cancer from which the patient has been disease-free for ≥ 3 years
* Patients with a known history of HIV seropositivity
* Active HCV infection (PCR + ; AST> 1.5-2x UN)
* Woman who is pregnant or breast feeding. Fertile patients not willing to use effective contraception during the study and 3 months after the end of treatment. Women of childbearing potential (WOCBP) are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months.
* Negative pregnancy test at baseline is required (serum β HCG).
* Male patient whose sexual partner(s) are WOCBP who are not willing to use a effective contraception during the study and 3 months after the end of treatment
* Nodular lymphocyte prevalence histological subtype

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2017-04-29 (Actual)

PRIMARY OUTCOMES:
Feasibility | After 4 dd-ABVD cycles (12 weeks after starting treatment)
  Proportion of patient with a dose intensity reduction (lower than 85% of planned dose)
Activity | After 2 dd-ABVD cycles (6 week after starting treatment)
  Percentage of FDG PET negativity after 2 dd-ABVD cycles will be considered as primary endpoints.

SECONDARY OUTCOMES:
Overall accuracy of each interim PET interpretation criteria after a minimum follow-up of three years | After 3 years of follow-up
  Concordance between pet results and patients prognosis
PFS | 2 years from the activation of therapy in the last patient enrolled onto the study.
  Progression free survival estimate (prognosis outcome)
OS | 2 years from the activation of therapy in the last patient enrolled onto the study.
  Overall survival estimate (prognosis outcome)
Toxicity | 2 years from the activation of therapy in the last patient enrolled onto the study.
  Proportion of early and late toxicities (G3/4 acute toxicities, secondary malignancies, cardiovascular and pulmonary events, infertility)
Predictive Value of each interim PET interpretation criteria after a minimum follow-up of three years | After 3 years of follow-up
  Concordance between pet results and patients prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, M.D., Principal Investigator — Humanitas Cancer Center - Department of Medical Oncology and Haematology
Locations (37):
- Italy (37):
  - UO Ematologia Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Dipartimento di Oncologia Medica ed Ematologia Istituto Clinico Humanitas, Rozzano, Milano
  - Oncologia HSR Giglio, Cefalù, Palermo
  - Oncologia Medica A Centro di Riferimento Oncologico, Aviano, Pordenone
  - U.O. Oncoematologia Ospedale "Andrea Tortora", Pagani, Salerno
  - UO Ematologia Ospedale San Donato, Arezzo
  - UO Ematologia con trapianto AOU Policlinico Consorziale, Bari
  - SOS Ematologia Divisione Medicina Interna Ospedale degli Infermi, Biella
  - Ematologia e CTMO Ospedale Businco, Cagliari
  - UOC Oncoematologia Garibaldi Nesima, Catania
  - UOC Ematologia Azienda Ospedaliera Cosenza, Cosenza
  - Unità Funzionale di Ematologia AOU Careggi, Florence
  - Ematologia- AOU San Martino IRCCS - IST, Genova
  - SC Medicina Trasfusionale ed Ematologia SS Ematologia ASLTO4, Ivrea
  - UO Ematologia PO Vito Fazzi, Lecce
  - IRST Meldola, Meldola
  - SC Ematologia AO Riuniti Papardo Piemonte, Messina
  - UO Oncoematologia AO San Carlo Borromeo Unità Semplice di Trapianto Midollo, Milan
  - Centro Oncoematologico Policlinico, Modena
  - Unità Complessa di Ematologia AO di Rilievo Nazionale A. Cardarelli, Napoli
  - SCDU Ematologia Università Piemonte Orientale, Novara
  - Oncoematologia e TMO Dopartimento Oncologia La Maddalena, Palermo
  - UO Complessa di Ematologia Ospedale di Parma, Parma
  - Clinica Ematologica Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ematologia Ospedale Santo Spirito, Pescara
  - UO Ematologia Ospedale Santa Maria delle Croci, Ravenna
  - SC Ematologia Azienda Ospedaliera Arcispedale Santa Maria Nuova, Reggio Emilia
  - UO Oncoematologia AUSL Rimini Ospedale Infermi, Rimini
  - Ematologia e Trapianto Istituto Regina Elena IFO, Roma
  - Ematologia Ospedale Sant'Andrea, Roma
  - Ematologia Università La Sapienza, Roma
  - Ematologia e Trapianti AO San Giovanni di Dio e Ruggi D'Aragona, Salerno
  - Azienda Ospedaliera Università Senese Clinica Ematologica Policlinico Le Scotte, Siena
  - Oncoematologia Università Perugia sede Terni, Terni
  - SC Ematologia AO Città della Salute e della Scienza, Torino
  - Clinica Ematologica AO S. Maria della Misericordia, Udine
  - UOC Ematologia Ospedale di Circolo, Varese

REFERENCES:
- [Derived] Santoro A, Mazza R, Spina M, Califano C, Specchia G, Carella M, Consoli U, Palombi F, Musso M, Pulsoni A, Kovalchuk S, Bonfichi M, Ricci F, Fabbri A, Liberati AM, Rodari M, Giordano L, Chimienti E, Balzarotti M, Sorasio R, Gallamini A, Ghiggi C, Ciammella P, Ricardi U, Chauvie S, Carlo-Stella C, Merli F. Dose-dense ABVD as first-line therapy in early-stage unfavorable Hodgkin lymphoma: results of a prospective, multicenter double-step phase II study by Fondazione Italiana Linfomi. Ann Hematol. 2021 Oct;100(10):2547-2556. doi: 10.1007/s00277-021-04604-x. Epub 2021 Jul 30. PMID 34327561